CLINICAL TRIAL: NCT03328949
Title: Prospective Multi-Center, Single Arm Post-Market Study (PMS) of the Shockwave Medical, Inc. Coronary Lithoplasty® System in Coronary Arteries
Brief Title: Shockwave Coronary Lithoplasty® Study (Disrupt CAD II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP61774
Record Dates: First submitted 2017-10-27; First posted 2017-11-01 (Actual); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Intravascular Coronary Lithotripsy System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- IVL Coronary Lithotripsy System (Experimental): All enrolled patients will receive treatment from the IVL coronary lithotripsy system prior to coronary stent placement.
  Interventions: Device: IVL Coronary Lithotripsy System

INTERVENTIONS:
Device: IVL Coronary Lithotripsy System — The coronary intravascular lithotripsy catheter is similar to other balloon devices that are routinely used during angioplasty procedures; however, it has electrodes inside the balloon which are designed to deliver energy to crack the calcified blockage using lithotripsy (acoustic energy).

SUMMARY:
The objective of this post market study is to examine the safety and performance of the Shockwave Coronary Intravascular Lithotripsy System for the treatment of narrowed coronary arteries before the doctor places a stent.

DETAILED DESCRIPTION:
The study will be conducted at 15 sites in Europe and up to 120 participants will be followed for 30 days post procedure.

Patients ≥18 years of age scheduled for stent procedure with evidence of significant calcified stenosis of left main, or left anterior descending, right coronary artery or left circumflex will be eligible to enroll in the study. The primary endpoint of the study will evaluate major adverse cardiac events post procedure including 1) cardiac related death, 2) heart attack, and 3) intervention to treat the coronary artery that was previously treated at the procedure visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years of age
2. Troponin must be less than or equal to the upper limit of lab normal value within 24 hours prior to the procedure OR if troponin is elevated, concomitant CK must be normal
3. The target vessel must have a TIMI flow 3 at baseline
4. Patients with significant (≥ 50% diameter stenosis) native coronary artery disease including stable or unstable angina and silent ischemia, suitable for PCI
5. Ability to tolerate dual antiplatelet agent (i.e. aspirin, clopidogrel, prasugrel, or ticagrelor) for 1 year and single antiplatelet therapy for life
6. Single lesion stenosis of protected LMCA, or LAD, RCA or LCX artery ≥50% in a reference vessel of 2.5 mm - 4.0 mm diameter and ≤ 32 mm length
7. Presence of calcification within the lesion on both sides of the vessel as assessed by angiography
8. Planned treatment of single lesion in one vessel
9. Ability to pass a 0.014" guide wire across the lesion
10. Patient, or authorized representative, signs a written Informed Consent form to participate in the study, prior to any study-mandated procedures
11. Patient is able and willing to comply with all assessments in the study

Exclusion Criteria:

1. Concomitant use of Atherectomy, Specialty balloon, or investigational coronary devices
2. Prior PCI procedure within the last 30 days of the index procedure
3. Patient has planned cardiovascular interventions within 30 days post index procedure
4. Second lesion with ≥50% stenosis in the same target vessel
5. Left ventricular ejection fraction < 40%
6. Patient refusing or not a candidate for emergency coronary artery bypass grafting (CABG) surgery
7. Uncontrolled severe hypertension (systolic BP >180 mm Hg or diastolic BP >110 mm Hg)
8. Severe renal failure with serum creatinine >2.5 mg/dL, unless on chronic dialysis
9. Untreated pre-procedural hemoglobin <10 g/dL
10. Coagulopathy manifested by platelet count <100,000 or International Normalized ratio (INR) >1.7 (INR is only required in patients who have taken warfarin within 2 weeks of enrollment)
11. Patients in cardiogenic shock
12. Acute myocardial infarction (MI) within the past one (1) month, and/or signs of active myocardial ischemia at the time of enrollment including elevated Troponin-I or T (with concomitant elevation of CK), ischemic ECG changes or chest pain
13. History of a stroke or transient ischemic attack (TIA) within 3 months
14. NYHA class III or IV heart failure
15. Active peptic ulcer or upper gastrointestinal (GI) bleeding within 6 months
16. Patients with a life expectancy of less than 1 year
17. Target vessel < 2.4 mm in diameter
18. Target lesion > 32 mm in length
19. Chronic Total Occlusion (CTO)
20. Previous stent procedure within 5 mm of target lesion
21. Angiographic evidence of a target lesion severe dissection prior to Coronary Lithoplasty treatment
22. Unprotected Left Main diameter stenosis ≥ 50%
23. Visible thrombus (by angiography) at target lesion site
24. Target lesion is located in a native vessel distal to anastomosis with a saphenous vein graft or LIMA/RIMA bypass
25. Patient has active systemic infection
26. Patient has connective tissue disease (e.g., Marfan's syndrome)
27. Patient has a hypercoagulable disorder
28. Uncontrolled insulin dependent diabetes
29. Patient has allergy to imaging contrast media for which they cannot be pre-medicated
30. Evidence of aneurysm in target vessel
31. Patient is pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Fajadet, MD, Principal Investigator — Clinic Pasteur; Carlo DiMario, MD, Principal Investigator — University of Florence
Locations (15):
- Onze-Lieve-Vrouwziekenhuis, Aalst, Belgium
- Aarhus Universitetshospital, Aarhus, Denmark
- France (2):
  - Institut Hospitalier Jacques Cartier, Massy
  - Clinique Pasteur, Toulouse
- Germany (3):
  - Universitaets-Herzzentrum Freiburg- Bad Krozingen, Bad Krozingen
  - Universitaetsklinikum Bonn, Bonn
  - UKGM Universitaetsklinikum Giessen, Giessen
- Italy (2):
  - AOU Careggi SOD Interventistica, Florence
  - San Raffaelle Hospital, Milan
- Netherlands (2):
  - Thorax Center, Erasmus MC, Rotterdam
  - Isala Zeikenhuis- Hartecentrum, Zwolle
- Hospital Universitario San Carlos, Madrid, Spain
- Uppsala University Hospital, Uppsala, Sweden
- United Kingdom (2):
  - King's College Hospital, London
  - Oxford University Hospitals, John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kereiakes DJ, Di Mario C, Riley RF, Fajadet J, Shlofmitz RA, Saito S, Ali ZA, Klein AJ, Price MJ, Hill JM, Stone GW. Intravascular Lithotripsy for Treatment of Calcified Coronary Lesions: Patient-Level Pooled Analysis of the Disrupt CAD Studies. JACC Cardiovasc Interv. 2021 Jun 28;14(12):1337-1348. doi: 10.1016/j.jcin.2021.04.015. Epub 2021 May 3. PMID 33939604
- [Derived] Ali ZA, Nef H, Escaned J, Werner N, Banning AP, Hill JM, De Bruyne B, Montorfano M, Lefevre T, Stone GW, Crowley A, Matsumura M, Maehara A, Lansky AJ, Fajadet J, Di Mario C. Safety and Effectiveness of Coronary Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Stenoses: The Disrupt CAD II Study. Circ Cardiovasc Interv. 2019 Oct;12(10):e008434. doi: 10.1161/CIRCINTERVENTIONS.119.008434. Epub 2019 Sep 25. PMID 31553205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment and enrollment took place at 15 clinical sites in 9 European countries between May 2018 and March 2019. A total of 120 subjects with calcified, stenotic de novo coronary arteries were enrolled and treated with the Coronary Intravascular Lithotripsy (IVL) System.
Groups:
- Coronary Intravascular Lithotripsy (IVL) System: All enrolled patients will receive treatment from the coronary intravascular lithotripsy (IVL) system prior to coronary stent placement.
  Coronary Intravascular Lithotripsy (IVL) System: The coronary intravascular lithotripsy catheter is similar to other balloon devices that are routinely used during angioplasty procedures; however, it has electrodes inside the balloon which are designed to deliver energy to crack the calcified blockage using lithotripsy (acoustic energy).
Period: Overall Study
Arm/Group | Coronary Intravascular Lithotripsy (IVL) System
Started | 120
Completed | 120
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Coronary Intravascular Lithotripsy (IVL) System
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 94
  More than one race | 2
  Unknown or Not Reported | 21
Region of Enrollment [Number; unit: participants]
  Netherlands | 4
  Sweden | 1
  Belgium | 9
  Denmark | 1
  Italy | 25
  United Kingdom | 19
  France | 19
  Germany | 29
  Spain | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With In-hospital Major Adverse Cardiac Events (MACE)
Description: The primary endpoint is the frequency of in-hospital major adverse cardiac events (MACE). MACE is defined as the following:
  * Cardiac death
  * Myocardial Infarction - defined as a CK-MB level > 3 times the upper limit of lab normal (ULN) value with or without new pathologic Q wave
  * TVR - defined as revascularization at the target vessel (inclusive of the target lesion) after the completion of the index procedure
Time Frame: Post-procedure through hospital discharge
Population: No imputation of or adjustments for missing data were performed for the primary analysis. The population for all analysis was the Intent-To-Treat (ITT) analysis set. ITT was defined as those subjects who had insertion of the IVL catheter attempted, defined as the point of enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Intravascular Lithotripsy (IVL) System
Number analyzed (Participants) | 120
Participants | 7

2. Secondary Outcome: Number of Participants With Clinical Success
Description: Performance will be assessed by the ability of the Lithotripsy System to produce acceptable residual stenosis (<50%) after stenting with no evidence of in-hospital MACE. Each patient that achieves both of these requirements will be considered a "clinical success", and the rate of clinical success among subjects will be evaluated.
Time Frame: During procedure through hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Intravascular Lithotripsy (IVL) System
Number analyzed (Participants) | 120
Participants | 120

3. Secondary Outcome: Number of Participants With Angiographic Success
Description: Angiographic success defined as success in facilitating stent delivery with <50% residual stenosis and without serious angiographic complications. Serious angiographic complications defined as severe dissection (Type D to F), perforation, abrupt closure, and persistent slow flow or persistent no reflow.
Time Frame: During procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Intravascular Lithotripsy (IVL) System
Number analyzed (Participants) | 120
Participants | 120

4. Secondary Outcome: Number of Participants Which Experienced Cardiac Death
Description: Number of patients who experienced a cardiac death at 30 days post-procedure.
Time Frame: 30 days post-procedure
Measure: Count of Participants; unit: Participants
Groups:
- Coronary Intravascular Lithotripsy (IVL) System: All enrolled patients will receive treatment from the IVL coronary lithotripsy system prior to coronary stent placement.
  Coronary Intravascular Lithotripsy (IVL) System: The coronary intravascular lithotripsy catheter is similar to other balloon devices that are routinely used during angioplasty procedures; however, it has electrodes inside the balloon which are designed to deliver energy to crack the calcified blockage using lithotripsy (acoustic energy).
Arm/Group | Coronary Intravascular Lithotripsy (IVL) System
Number analyzed (Participants) | 120
Participants | 1

ADVERSE EVENTS:
Time Frame: From time of enrollment through 30 days
Arm/Group | Coronary Intravascular Lithotripsy (IVL) System
All-Cause Mortality (participants affected / at risk) | 1/120
Serious Adverse Events (participants affected / at risk) | 13/120
Other Adverse Events (participants affected / at risk) | 29/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coronary Intravascular Lithotripsy (IVL) System (N=120)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Arrhythmia (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Coronary artery dissection (Cardiac disorders) | 3 (3)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Paroxysmal atrioventricular block (Cardiac disorders) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Myocardial necrosis marker increased (Investigations) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coronary Intravascular Lithotripsy (IVL) System (N=120)
Angina pectoris (Cardiac disorders) | 2 (2)
Coronary artery dissection (Cardiac disorders) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 3 (3)
Vascular access site pain (Injury, poisoning and procedural complications) | 2 (2)
Myocardial necrosis marker increased (Investigations) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Macule (Skin and subcutaneous tissue disorders) | 1 (1)
Haemodynamic instability (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After publication of the multi-center Study, or earlier with Sponsor's prior written consent, the Institution may publish the results of its subjects enrolled in the Study after first complying with this Section 9 of the contract. The Institution agrees to submit any proposed publications to Sponsor for review and comment at least forty-five (45) days in advance of submitting such proposed publications to a publisher or other third party.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT03328949/Prot_SAP_000.pdf